CLINICAL TRIAL: NCT01875796
Title: Integrated CBT for Cannabis Dependence With Co-occurring Anxiety Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Julia Buckner, Associate Professor, Louisiana State University and A&M College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDA031937A; 1R34DA031937-01 (NIH)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Cannabis Dependence; Anxiety Disorders; Cannabis Use Disorder; Cannabis Abuse
Keywords: cannabis; marijuana; anxiety; transdiagnostic; dual diagnosis; cannabis abuse; cannabis dependence; cannabis use disorder
MeSH Terms: conditions — Marijuana Abuse; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cannabis & Anxiety Reduction Treatment (Experimental): Cognitive-behavioral treatment program that integrates strategies to manage both cannabis use and anxiety with techniques to address motivation to change cannabis use.
  Interventions: Behavioral: Cognitive-Behavioral Therapy; Behavioral: Motivation Enhancement Therapy; Behavioral: Integrated Cannabis and Anxiety Reduction Treatment; Behavioral: False Safety Behavior Elimination Therapy
- Motivation/cognitive-behavioral therapy (Active Comparator): Motivational Enhancement Therapy (MET) and cognitive-behavioral therapy (CBT) that includes techniques to address motivation to change cannabis use with strategies to manage use.
  Interventions: Behavioral: Cognitive-Behavioral Therapy; Behavioral: Motivation Enhancement Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy
Behavioral: Motivation Enhancement Therapy
Behavioral: Integrated Cannabis and Anxiety Reduction Treatment
  Arms: Cannabis & Anxiety Reduction Treatment
Behavioral: False Safety Behavior Elimination Therapy
  Other Names: Transdiagnostic anxiety disorder treatment
  Arms: Cannabis & Anxiety Reduction Treatment

SUMMARY:
This project tests the feasibility and utility of a novel, integrated approach to treatment of patients with cannabis use disorder (CUD) and anxiety disorders.

DETAILED DESCRIPTION:
Cannabis use disorder (CUD) is the most common illicit substance dependence and people with CUD are highly vulnerable to anxiety disorders. The co-occurrence of anxiety disorders among those with CUD is a pressing public health matter given elevated anxiety is related to poorer cannabis treatment outcomes. Cannabis-related problems among those with anxiety disorders may be maintained by a reliance on cannabis to manage anxiety. Investigations of the treatment of these conditions when they co-occur have been virtually absent. Motivation enhancement therapy (MET) combined with cognitive-behavioral therapy (CBT) is an efficacious intervention for cannabis CUD, yet outcomes are highly limited for anxious patients. Transdiagnostic anxiety treatments can facilitate the treatment of patients with anxiety psychopathology regardless of the specific type of anxiety disorder. One such treatment, False Safety Behavior Elimination Treatment (FSET), may be particularly useful with anxious patients with CUD as it focuses on the elimination of behaviors that may be effective in decreasing anxiety in the short-term, but can maintain and even exacerbate anxiety in the long-term (i.e., false safety behaviors). The use of cannabis to manage anxiety can, therefore, be targeted in such a treatment. This project tests the feasibility and utility of a novel, integrated approach to treatment of patients with CUD and anxiety disorders. Phase I of the project includes development and refinement of a specialized group protocol (i.e., Integrated Cannabis and Anxiety Reduction Treatment or ICART) for integrating MET-CBT for CUD with FSET. The initial protocol will be modified based on the experience gained during group treatment with the integrated treatment. Phase II will be a randomized controlled trial examining the relative efficacy of the refined ICART treatment versus MET-CBT alone. After post-treatment assessments, the ICART group will be followed for 3 months to examine maintenance of gains; the participants originally assigned to the control condition will be offered ICART. It is hypothesized that ICART will produce better outcomes than the control.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cannabis use disorder
2. An additional diagnosis of an anxiety disorder
3. Patient reports that at least some of his/her cannabis use is aimed at reducing anxiety and/or for social facilitation.
4. Patient reports that cannabis is his/her substance of choice for anxiety management.
5. Concurrent use of psychotropic medications (e.g., selective serotonin reuptake inhibitors) is permitted as long as patients have been on a stable dose for at least three months prior to entering the study and they are willing to remain stable on their medication for the duration of treatment.
6. Age between 18 and 65 years.
7. English language fluency.
8. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Alcohol or illicit substance (non-cannabis) dependence.
2. Cannabis use behavior sufficiently uncontrolled that proper participation in study protocol would likely be disrupted.
3. History of schizophrenia, bipolar disorder, or organic brain syndrome.
4. Prominent suicidal ideation with intent that is judged to be clinically significant.
5. Mental retardation or another pervasive developmental disability (e.g., Asperger's Disorder).
6. Sufficiently socially unstable as to preclude completion of study requirements (e.g., homeless).
7. Prior simultaneous cognitive behavioral treatment for cannabis dependence and anxiety disorders.
8. Legally mandated to receive substance abuse treatment.
9. Report of current participation in or intent to participate in an additional (i.e., treatments other than MET-CBT or MET alone) anxiety or substance abuse treatment method during the course of the study.
10. Unwilling to maintain stable dose of regularly-dosed medications during the study
11. Unwilling to cease PRN (pro re nata or "as needed") use of benzodiazepines or other fast-acting anxiolytics prior to entrance into social situations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
cannabis use | change from baseline to weeks 6, 12, & 32
cannabis-related problems | change from baseline to weeks 6, 12, & 32

SECONDARY OUTCOMES:
anxiety | change from baseline to weeks 6, 12, & 32

CONTACTS AND LOCATIONS:
Overall Officials: Julia D Buckner, PhD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans; Michael J Zvolensky, PhD, Principal Investigator — University of Houston
Locations (1):
- Louisiana State University Anxiety & Addictive Behaviors Clinic, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Buckner JD, Morris PE, Zvolensky MJ. Integrated cognitive-behavioral therapy for comorbid cannabis use and anxiety disorders: The impact of severity of cannabis use. Exp Clin Psychopharmacol. 2021 Jun;29(3):272-278. doi: 10.1037/pha0000456. Epub 2021 Apr 22. PMID 34264732